CLINICAL TRIAL: NCT06141083
Title: Effect of TCI188 Probiotic on Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N202307006
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Periodontal Diseases
Keywords: Pediococcus acidilactici; Probiotics
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo chewable tablets (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- TCI188 Probiotic chewable tablets (Experimental)
  Interventions: Dietary Supplement: TCI188 Probiotic

INTERVENTIONS:
Dietary Supplement: TCI188 Probiotic — take two tablets per day
  Other Names: Pediococcus acidilactici TCI188
  Arms: TCI188 Probiotic chewable tablets
Dietary Supplement: Placebo — take two tablets per day
  Arms: Placebo chewable tablets

SUMMARY:
To assess the efficacy of TCI188 (Pediococcus acidilactici) Probiotic on Oral Health

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old
* Participants suffer from severe periodontal disease throughout the mouth with symptoms at third and fourth stages, do not have immediate indications for the extraction of multiple teeth or complex denture stimulation, and have not undergone periodontal planing within one year.

Exclusion Criteria:

* Participants have had periodontal or antimicrobial treatment within the past 6 months
* Participants are smokers, pregnant or with systemic diseases
* Participants had probiotic supplements or with history of adverse reactions to lactose or fermented dairy products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
The change of clinical oral measurements- Probing pocket depth (PPD) | before root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  The values of Probing pocket depth (PPD) was utilized to evaluate oral status.
The change of clinical oral measurements- Bleeding on probing (BOP) | before root planning, after root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  The values of Bleeding on probing (BOP) was utilized to evaluate oral status.

SECONDARY OUTCOMES:
The change of clinical oral measurements- Plaque index (PI) | before root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  The values of Plaque index (PI) was utilized to evaluate oral status.
The change of clinical oral measurements- Clinical attachment level (CAL) | before root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  The values of Clinical attachment level (CAL) was utilized to evaluate oral status.
The change of clinical oral measurements- Gingival index (GI) | before root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  The values of Gingival index (GI) was utilized to evaluate oral status.
The change of inflammatory markers (IL-10, IL-1beta) of saliva | before root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  The levels of interleukin-10 (IL-10), interleukin-1beta (IL-1beta) in saliva were utilized to evaluate oral inflammation status.
The change of oral microflora | before root planning, after root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  The relative abundance of Streptococcus mutans, Porphyromonas gingivalis, Streptococcus salivarius, Pediococcus acidilactici were utilized to evaluate the change of oral microflora.
The change of liver function biomarkers (AST, ALT) of blood | before root planning, after root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  Fasting venous blood was sampled to measure liver function biomarkers- Aspartate Transaminase (AST), Alanine aminotransferase (ALT), Blood urea nitrogen (BUN), Creatinine, High-sensitivity CRP (Hs-CRP), Interleukin.
The change of renal function biomarkers (BUN, CRE) of blood | before root planning, after root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  Fasting venous blood was sampled to measure renal function biomarkers- Blood urea nitrogen (BUN), Creatinine (CRE).
The change of inflammatory biomarkers (Hs-CRP, IL-10, IL-1beta) of blood | before root planning, after root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  Fasting venous blood was sampled to measure inflammatory biomarkers- High-sensitivity CRP (Hs-CRP), Interleukin-10 (IL-10), Interleukin-1beta(IL-1beta).
The change of Bad breath | before root planning, after root planning, after taking chewable tablets for 6-8 weeks, and after finishing taking chewable tablets for 12 weeks
  The Bad Breath Tester was utilized to measure Bad breath. The Bad breath detection level is 0~5.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Wei Wang, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan, Taiwan